CLINICAL TRIAL: NCT02933645
Title: Effects of Intranasal Insulin Administration on Tissue Specific Insulin Sensitivity
Acronym: NASO-PET
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Turku University Hospital (Other Government)
Collaborators: University Hospital Tuebingen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Basic Science
Other Study IDs: T210/2015; 2015-005392-24 (EudraCT Number)
Record Dates: First submitted 2016-05-11; First posted 2016-10-14 (Estimated); Last update posted 2018-01-26 (Actual); Status verified 2018-01

CONDITIONS: Insulin Resistance
Keywords: Insulin; Intranasal; Glucose/metabolism; Glucose homeostasis
MeSH Terms: conditions — Insulin Resistance | interventions — Insulin; Insulin Aspart; Insulin Detemir

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Insulin nasal spray (Active Comparator): Subjects administer 2 intranasal sprays into each nostril every minute for 4 minutes, a total of 16 sprays. Sprays contain fast-acting human insulin Actrapid (Novo Nordisk A/S, Bagsvaerd, Denmark). The glass spray flasks are produced by AeroPump GmBH, Germany and give 0,1 ml of fluid per spray. To account for the small amount of insulin absorbed into circulation after the insulin nasal sprays, on the placebo day subjects will be administered 2.5 mU/kg of additional intravenous insulin (Actrapid, Novo Nordisk A/S, Bagsvaerd, Denmark) over 15 minutes.
  30 min before spray administration a hyperinsulinemic euglycemic clamp will be started and continued for 170 minutes. 40 min after spray administration [18F]-FDG PET-CT scan lasting 100 min is started.
  Interventions: Drug: Actrapid; Radiation: [18F]-FDG PET-CT; Drug: Hyperinsulinemic euglycemic clamp
- Placebo nasal spray (Placebo Comparator): Subjects administer 2 intranasal sprays into each nostril every minute for 4 minutes, a total of 16 sprays. Sprays contain Insulin Diluting Medium for Novorapid and Levemir (Novo Nordisk A/S, Bagsvaerd,Denmark). The glass spray flasks are produced by AeroPump GmBH, Germany and give 0,1 ml of fluid per spray. To account for the small amount of insulin absorbed into circulation after the insulin nasal sprays, on the placebo day subjects will be administered 2.5 mU/kg of additional intravenous insulin (Actrapid, Novo Nordisk A/S, Bagsvaerd,Denmark) over 15 min.
  30 min before spray administration a hyperinsulinemic euglycemic clamp will be started and continued for 170 minutes. 40 min after spray administration [18F]-FDG PET-CT scan lasting 100 min is started.
  Interventions: Drug: Placebo; Radiation: [18F]-FDG PET-CT; Drug: Hyperinsulinemic euglycemic clamp

INTERVENTIONS:
Drug: Actrapid — Subjects administer 2 intranasal sprays into each nostril every minute for 4 minutes, a total of 16 sprays or 160 IU of fast-acting human insulin (Actrapid, Novo Nordisk A/S, Bagsvaerd, Denmark). The glass spray flasks are produced by AeroPump GmBH, Germany and give 0,1 ml of fluid per spray.
  Other Names: ATC-code A10AB01
  Arms: Insulin nasal spray
Drug: Placebo — Subjects administer 2 intranasal sprays into each nostril every minute for 4 minutes, a total of 16 sprays. Sprays contain Insulin Diluting Medium for Novorapid and Levemir (Novo Nordisk A/S, Bagsvaerd, Denmark). The glass spray flasks are produced by AeroPump GmBH, Germany and give 0,1 ml of fluid per spray. To account for the small amount of insulin absorbed into circulation after the insulin nasal sprays, on the placebo day subjects will be administered 2.5 mU/kg of additional intravenous insulin (Actrapid, Novo Nordisk A/S, Bagsvaerd, Denmark) over 15 minutes.
  Other Names: Insulin Diluting Medium for Novorapid and Levemir
  Arms: Placebo nasal spray
Radiation: [18F]-FDG PET-CT — All subjects will undergo two positron emission tomography (PET) studies. On both visits they are injected with 185 MBq [18F]-fluorodeoxyglucose and scanned with a combined PET and computed tomography scanner.
  Other Names: Tissue specific insulin sensitivity measurement
Drug: Hyperinsulinemic euglycemic clamp — All subjects will undergo two hyperinsulinemic euglycemic clamp studies. The insulin infusion will be administered intravenously at a steady rate of 0.25 mU/kg/min for approximately 170 minutes. Glucose will be administered intravenously as a 200 mg/ml fluid to at varying rate to maintain euglycemia.
  Other Names: Whole-body insulin sensitivity measurement

SUMMARY:
Recent research has suggested that intranasally administered insulin can reach the brain quickly without passing through circulation and evoke increased insulin sensitivity and tissue glucose consumption during insulin stimulation (low-dose hyperinsulinemic, euglycemic clamp). It is still not known what mechanism causes these changes or what tissues are involved in this.

In this study, the changes in tissue-specific insulin sensitivity and glucose uptake will be investigated by using glucose-analogue radiotracer ([18F]-fluorodeoxyglucose) with positron emission tomography (PET) imaging during insulin stimulation. Ten healthy males are studied, each receiving nasal sprays containing insulin or placebo in a randomized order on two separate days. After spray administration, glucose uptake in skeletal muscle, liver, subcutaneous and visceral adipose tissue, myocardium, intestines, brown adipose tissue and brain assessed by PET imaging and glucose uptake in these tissues is analyzed. Endogenous glucose production is calculated facilitating the measurements glucose and radiotracer uptake in tissues and tracer loss into urine.

As skeletal muscle consumes most of the glucose available, it is likely that administration of insulin sprays will result in an increased uptake in this tissue. Some increase in glucose uptake might also be seen in other tissue types after insulin spray versus placebo spray administration.

DETAILED DESCRIPTION:
The objective of this study is to investigate the effects of intranasally administered insulin versus placebo on tissue specific glucose uptake of the key metabolic organs as well as on endogenous glucose production.

SAMPLE SIZE:

A total of ten (n=10) healthy males are planned to be included, and the study is conducted with a cross-over design with each subject being investigated twice, once using intranasal insulin and once using intranasal placebo in single-blinded randomized order.

SCREENING VISIT/ELIGIBILITY:

Main inclusion and exclusion criteria will be evaluated at a screening visit. This visit will include a frequently-sampled 75 g oral glucose tolerance test as well as anthropometric measurements and clinical examination.

PET STUDY VISITS:

On the PET study days two cannulas will be inserted, one in a radial or an antecubital vein for tracer injection and infusion of glucose and insulin, another in the opposite radial or antecubital vein for blood sampling. The arm where the samples are taken will be kept warm to obtain arterialized venous blood. The subjects will rest in supine position on the PET/CT scanner bed during the study.

HYPERINSULINEMIC EUGLYCEMIC CLAMP:

Whole-body insulin sensitivity will be assessed by hyperinsulinemic euglycemic clamp with an primed insulin infusion rate of 0.25 mU/kg/min. To maintain the glucose level at 5.0 mmol/l intravenous glucose infusion is administered individually as needed to maintain euglycemia.

NASAL SPRAY ADMINISTRATION:

After 30 minutes of intravenous insulin infusion, the subjects will receive either 160 IU human insulin or placebo intranasally. The small amount of insulin known to be absorbed into circulation after the insulin nasal spray will be mimicked on placebo day. Therefore subjects will be administered 2.5 mU/kg of additional intravenous insulin over 15 minutes together with placebo spray administration.

LABORATORY SAMPLES:

To verify comparable insulin levels in circulation during the study, serum insulin and C-peptide levels will be determined in fasting state, and repeatedly throughout the experiment.

BLINDING:

The clinician and the study nurse are aware which spray is given, but subjects are blinded and additional insulin infusion on placebo day is done in a manner that the subjects remain blinded. The sprays are given on a randomized order. The randomization code was generated by a statistician using SAS, version 9.3 for Windows. The randomization block size was four and the method was permuted block randomization. The randomization was done for 16 subjects in case of discontinuations.

HEART RATE VARIABILITY:

Heart rate variability is recorded to evaluate changes in autonomous nervous system activity after spray administration on both visits. Polar RS800CX heart rate monitor (Polar Electro Ltd., Kempele, Finland) with two electrodes is used.

FDG-PET-IMAGING:

70 minutes after the start of clamp and 40 minutes after the application of nasal sprays the positron emission tomography (PET) scanning is started with the injection of glucose-analogue tracer labeled with positron-emitting fluorine-18 ([18F]-fluorodeoxyglucose, [18F]-FDG). PET/CT, GE DiscoveryTM ST System (General Electric Medical Systems, Milwaukee, WI, USA) with final resolution of 3.75 mm in PET images is used. All data will be corrected for dead-time, decay and measured photon attenuation. Dynamic PET-scans will be reconstructed with iterative reconstruction method. Radiotracer [18F]-FDG is produced in the PET Centre radiochemistry laboratory. Plasma radioactivity is measured with an automatic gamma counter by a medical technologist in the laboratory of the Turku PET Centre (Wizard 1480 3", Wallac, Turku, Finland).

PET-IMAGE ANALYSIS:

To determine tissue-specific glucose uptake during insulin stimulation from PET data, time-activity-curves of tissue activity and activity measured from plasma during the scanning are analysed graphically to define tracer's fractional uptake (Ki). To calculate glucose uptake rate (reported as µmol/kg/min), Ki is multiplied with plasma glucose level, divided with a constant that accounts for the differences in transport and dephosphorylation rates between D-glucose and FDG (lumped constant, LC) and divided with tissue specific gravity. Based on previous studies the LC is 1,2 for skeletal muscle; 1,0 for heart and liver; 1,14 for adipose tissue; 1,1 for intestines and 0,8 for brain. After the PET/CT an urine sample will be collected to quantify endogenous glucose production (EGP). This will be determined by subtracting urine loss and glucose infusion rate from rate of glucose disappearance.

ELIGIBILITY:
Inclusion Criteria:

1. BMI 18,5-25 kg/m2
2. Fasting plasma glucose less than 6.1 mmol/l
3. Normal 2-hour oral glucose tolerance test (OGTT)

Exclusion Criteria:

1. Any chronic disease or medication that could affect glucose metabolism
2. History of anorexia nervosa or bulimia
3. Smoking of tobacco, taking of snuffs, or use of narcotics
4. Abusive use of alcohol
5. Any other condition that in the opinion of the investigator could create a hazard to the subject safety, endanger the study procedures or interfere with the interpretation of study results

Ages: 20 Years to 35 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 10 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2016-12 (Actual); Study Completion 2016-12 (Actual)

PRIMARY OUTCOMES:
Skeletal muscle glucose uptake | Data is collected during 100 min PET scan started 40 min after spray administration.
  Change in skeletal muscle insulin stimulated glucose uptake (μmol/min/kg) after insulin versus placebo nasal spray administration.

SECONDARY OUTCOMES:
Endogenous glucose production | Data is collected during 100 min PET scan started 40 min after spray administration.
  Change in endogenous glucose production after insulin versus placebo nasal spray administration (μmol/min/kg) . Endogenous glucose production is determined by subtracting urine loss and glucose infusion rate from rate of glucose disappearance facilitating measurements of fluorodeoxyglucose concentrations in plasma after the injection and in urine right after the end of PET scanning.
Liver glucose uptake | Data is collected during 100 min PET scan started 40 min after spray administration.
  Change in liver insulin stimulated glucose uptake (μmol/min/kg) after insulin versus placebo nasal spray administration.

CONTACTS AND LOCATIONS:
Overall Officials: Pirjo Nuutila, MD,PhD, Principal Investigator — Turku University Hospital
Locations (1):
- Turku PET Centre, Turku, Finland

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Heni M, Wagner R, Kullmann S, Veit R, Mat Husin H, Linder K, Benkendorff C, Peter A, Stefan N, Haring HU, Preissl H, Fritsche A. Central insulin administration improves whole-body insulin sensitivity via hypothalamus and parasympathetic outputs in men. Diabetes. 2014 Dec;63(12):4083-8. doi: 10.2337/db14-0477. Epub 2014 Jul 15. PMID 25028522
- [Background] Heni M, Kullmann S, Preissl H, Fritsche A, Haring HU. Impaired insulin action in the human brain: causes and metabolic consequences. Nat Rev Endocrinol. 2015 Dec;11(12):701-11. doi: 10.1038/nrendo.2015.173. Epub 2015 Oct 13. PMID 26460339
- [Background] Born J, Lange T, Kern W, McGregor GP, Bickel U, Fehm HL. Sniffing neuropeptides: a transnasal approach to the human brain. Nat Neurosci. 2002 Jun;5(6):514-6. doi: 10.1038/nn849. No abstract available. PMID 11992114
- [Background] DeFronzo RA, Tobin JD, Andres R. Glucose clamp technique: a method for quantifying insulin secretion and resistance. Am J Physiol. 1979 Sep;237(3):E214-23. doi: 10.1152/ajpendo.1979.237.3.E214. PMID 382871
- [Background] Patlak CS, Blasberg RG. Graphical evaluation of blood-to-brain transfer constants from multiple-time uptake data. Generalizations. J Cereb Blood Flow Metab. 1985 Dec;5(4):584-90. doi: 10.1038/jcbfm.1985.87. PMID 4055928
- [Background] Peltoniemi P, Lonnroth P, Laine H, Oikonen V, Tolvanen T, Gronroos T, Strindberg L, Knuuti J, Nuutila P. Lumped constant for [(18)F]fluorodeoxyglucose in skeletal muscles of obese and nonobese humans. Am J Physiol Endocrinol Metab. 2000 Nov;279(5):E1122-30. doi: 10.1152/ajpendo.2000.279.5.E1122. PMID 11052968
- [Background] Botker HE, Bottcher M, Schmitz O, Gee A, Hansen SB, Cold GE, Nielsen TT, Gjedde A. Glucose uptake and lumped constant variability in normal human hearts determined with [18F]fluorodeoxyglucose. J Nucl Cardiol. 1997 Mar-Apr;4(2 Pt 1):125-32. doi: 10.1016/s1071-3581(97)90061-1. PMID 9115064
- [Background] Iozzo P, Jarvisalo MJ, Kiss J, Borra R, Naum GA, Viljanen A, Viljanen T, Gastaldelli A, Buzzigoli E, Guiducci L, Barsotti E, Savunen T, Knuuti J, Haaparanta-Solin M, Ferrannini E, Nuutila P. Quantification of liver glucose metabolism by positron emission tomography: validation study in pigs. Gastroenterology. 2007 Feb;132(2):531-42. doi: 10.1053/j.gastro.2006.12.040. Epub 2006 Dec 21. PMID 17258736
- [Background] Virtanen KA, Peltoniemi P, Marjamaki P, Asola M, Strindberg L, Parkkola R, Huupponen R, Knuuti J, Lonnroth P, Nuutila P. Human adipose tissue glucose uptake determined using [(18)F]-fluoro-deoxy-glucose ([(18)F]FDG) and PET in combination with microdialysis. Diabetologia. 2001 Dec;44(12):2171-9. doi: 10.1007/s001250100026. PMID 11793018
- [Background] Honka H, Makinen J, Hannukainen JC, Tarkia M, Oikonen V, Teras M, Fagerholm V, Ishizu T, Saraste A, Stark C, Vahasilta T, Salminen P, Kirjavainen A, Soinio M, Gastaldelli A, Knuuti J, Iozzo P, Nuutila P. Validation of [18F]fluorodeoxyglucose and positron emission tomography (PET) for the measurement of intestinal metabolism in pigs, and evidence of intestinal insulin resistance in patients with morbid obesity. Diabetologia. 2013 Apr;56(4):893-900. doi: 10.1007/s00125-012-2825-5. Epub 2013 Jan 20. PMID 23334481
- [Background] Wu HM, Bergsneider M, Glenn TC, Yeh E, Hovda DA, Phelps ME, Huang SC. Measurement of the global lumped constant for 2-deoxy-2-[18F]fluoro-D-glucose in normal human brain using [15O]water and 2-deoxy-2-[18F]fluoro-D-glucose positron emission tomography imaging. A method with validation based on multiple methodologies. Mol Imaging Biol. 2003 Jan-Feb;5(1):32-41. doi: 10.1016/s1536-1632(02)00122-1. PMID 14499160
- [Background] Iozzo P, Gastaldelli A, Jarvisalo MJ, Kiss J, Borra R, Buzzigoli E, Viljanen A, Naum G, Viljanen T, Oikonen V, Knuuti J, Savunen T, Salvadori PA, Ferrannini E, Nuutila P. 18F-FDG assessment of glucose disposal and production rates during fasting and insulin stimulation: a validation study. J Nucl Med. 2006 Jun;47(6):1016-22. PMID 16741312